CLINICAL TRIAL: NCT05393817
Title: Changes in Diaphragmatic Activity Before and After Caffeine Citrate Administration and Discontinuation
Brief Title: Caffeine Citrate Use and Electronic Activity of the Diaphragm (EDI) Changes
Status: Completed | Type: Observational
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Sook Kyung Yum, Professor, The Catholic University of Korea
Other Study IDs: KC22OISI0314
Record Dates: First submitted 2022-05-20; First posted 2022-05-26 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Preterm; Apnea of Prematurity; Caffeine
MeSH Terms: conditions — Premature Birth; Apnea | interventions — caffeine citrate; Caffeine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low-dose group: Infants receiving low dose caffeine citrate (up to 10mg/kg/day)
  Interventions: Drug: caffeine citrate
- High dose group: Infants receiving high dose caffeine citrate (exceeding 10mg/kg/day)
  Interventions: Drug: caffeine citrate

INTERVENTIONS:
Drug: caffeine citrate — caffeine citrate administration, dosage decided by the the physician on duty, within the range of routine management (5mg/kg/day ~ 20mg/kg/day)
  Other Names: caffeine; Neocaf injection [20mg] (Pharmbio Korea Inc.); Neocaf solution [20mg] (Pharmbio Korea Inc.)

SUMMARY:
Caffeine citrate, the first-line agent for apnea of prematurity, enhances diaphragmatic activity. EDI values of neurally adjusted ventilatory assist (NAVA) modes can be used to quantify the diaphragmatic activity triggered by electrical impulse from the respiratory center. This study aims to evaluate the EDI changes following caffeine citrate administration and cessation in preterm infants, and whether such changes are affected by different doses used variably in clinical settings.

DETAILED DESCRIPTION:
Caffeine citrate has been used as the first-line agent for apnea of prematurity. It works via mechanisms including stimulation of the respiratory center in medulla, increasing sensitivity to carbon dioxide retention, and increment in diaphragmatic activity. The effect of caffeine citrate has been evaluated largely based on parameters concerning clinical symptoms (e.g., decrease in the number of apnea, extubation success, decreased incidence of bronchopulmonary dysplasia) but not quantified parameters of actual diaphragmatic activity. Also, while usual doses of caffeine administration is described in the literature, consensus on the effect of caffeine citrate depending on different dosages has not been established.

The current study aims to evaluate effect of caffeine citrate by quantifying the electrical impulses of diaphragmatic activity using EDI values captured from neurally adjusted ventilatory assist (NAVA) mode.

Out of preterm infants necessitating invasive or non-invasive ventilators, those who are supported by invasive or non-invasive NAVA would be recruited. EDI changes would be monitored for the following timepoints: at the administration of caffeine citrate loading dose, 1st maintenance dose after loading, and at cessation of caffeine citrate.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born at less than 34 weeks' gestation who are supported by invasive or non-invasive NAVA

Exclusion Criteria:

* major congenital anomaly, chromosomal or genetic abnormality

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants admitted to the neonatal intensive care unit of the study site
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
EDI change after caffeine citrate loading dose | 20 minutes before ~ 20 minutes after loading dose of caffeine citrate
  changes in EDI min and EDI peak values (μV) after the loading dose administration
EDI change after caffeine citrate maintenance dose | 20 minutes before ~ 20 minutes after 1st maintenance dose of caffeine citrate
  changes in EDI min and EDI peak values (μV) after the 1st maintenance dose
EDI change after caffeine citrate cessation | 20 minutes before ~ 48 hours after caffeine citrate discontinuation (discontinuation time point definition: 48~96 hours after the last dose of caffeine citrate administration)
  changes in EDI min and EDI peak values (μV) after caffeine discontinuation

SECONDARY OUTCOMES:
short-term effect of caffeine citrate administration | 24 hours before ~ 24 hours after caffeine citrate administration
  number of apnea and/or bradycardia

OTHER OUTCOMES:
respiratory outcome of caffeine citrate administration (1) | During neonatal intensive care unit stay up to 48 weeks postmenstrual age (average of 3 months)
  duration of invasive mechanical ventilation (days)
respiratory outcome of caffeine citrate administration (2) | 36 weeks postmenstrual age or at discharge, whichever comes first
  bronchopulmonary dysplasia severity (no/mild/moderate/severe)

CONTACTS AND LOCATIONS:
Overall Officials: Sook Kyung Yum, MD, PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- Seoul St. Mary's Hospital, Seoul, Seocho-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No